CLINICAL TRIAL: NCT01735084
Title: Pneumococcal Conjugate Vaccine (PCV) Schedules for the Northern Territory (NT): Randomised Controlled Trial of Booster Vaccines to Broaden and Strengthen Protection From Invasive and Mucosal Infections.
Brief Title: Using Pneumococcal Vaccines in Combination for Maximum Protection From Ear and Lung Infections in First 3 Years of Life
Acronym: PREV-IX_B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1046999
Record Dates: First submitted 2012-11-15; First posted 2012-11-28 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Otitis Media; Febrile Illness; Cough; Lower Respiratory Tract Infection; Upper Respiratory Tract Infection
Keywords: randomized controlled trial; pneumococcal conjugate vaccines; booster dose; immunogenicity; nasopharyngeal carriage; Australian Indigenous; pediatric
MeSH Terms: conditions — Otitis Media; Cough; Respiratory Tract Infections | interventions — 13-valent pneumococcal vaccine; PHiD-CV vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prevenar13 (Experimental): The booster dose of Prevenar13 is 0.5 mL given intramuscularly only, with care to avoid injection into or near nerves and blood vessels. The preferred sites are anterolateral aspect of the thigh (vastus lateralis muscle) in infants or the deltoid muscle of the upper arm in young children.
  Interventions: Biological: Prevenar13
- Synflorix (Experimental): The booster vaccination schedule consists of one dose of 0.5 ml with an interval of at least 1 month between doses.
  Interventions: Biological: Synflorix

INTERVENTIONS:
Biological: Prevenar13 — The vaccine is a ready to use homogeneous white suspension for intramuscular injection, supplied as a pre-filled syringe.
  Active ingredients
  Each 0.5 mL dose contains:
  2.2 μg of pneumococcal purified capsular polysaccharides for serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F and 23F 4.4 μg of pneumococcal purified capsular polysaccharides for serotype 6B. Each serotype is individually conjugated to non-toxic diphtheria CRM197 protein and adsorbed on aluminium phosphate (0.565 mg).
  Other Names: PCV13; Prevnar13
  Arms: Prevenar13
Biological: Synflorix — The 10-valent vaccine contains 1 µg of purified capsular polysaccharide of pneumococcal serotypes 1, 5, 6B, 7F, 9V, 14, and 23F conjugated to protein D, 3 µg of serotype 4 conjugated to protein D, 3 µg of serotype 18C conjugated to tetanus toxoid and 3 µg of serotype 19F conjugated to diphtheria toxoid.
  Other Names: PHiD-CV; PHiD-CV10
  Arms: Synflorix

SUMMARY:
HYPOTHESES:

1. That infants receiving PHiD-CV10 as a booster at 12 months of age, compared to controls having no PHiD-CV10 booster (i.e. standard PCV13), will have higher HiD antibody levels, lower carriage of NTHi, and less tympanic membrane perforation at 18 and 36 months of age.
2. That infants receiving PCV13 as a booster at 12 months of age, compared to controls having no PCV13 (i.e. PHiD-CV10 booster) will have higher antibody levels to serotypes 3, 6A and 19A, less carriage of these serotypes, and less tympanic membrane perforation at 18 and 36 months of age.

DETAILED DESCRIPTION:
BACKGROUND:

PCV13 is now the recommended PCV in Australia, as 3+0 for non-Indigenous children and as 3+1 for Indigenous children in Western Australia, Queensland and Northern Territory. The decision to recommend PCV13 over PHiD-CV10 has been primarily driven by the increase in cases of invasive pneumococcal disease due to serotype 19A(1). However for the NT, in the last 3 years there has been one case of serotype 3, 6A or 19A invasive pneumococcal disease (IPD) per year in Indigenous children less than 2 years of age. By contrast, almost 20% of young Indigenous children have perforated tympanic membranes of which 60% are associated with NTHi, compared to 3% having serotypes 3, 6A or 19A.

The PREV-IX_COMBO trial is a randomised controlled trial (RCT) of these two pneumococcal conjugate vaccines currently licensed in Australia. Participating Indigenous infants living in remote communities in 4 regions of the NT are randomised between 28 and 38 days of age and allocated to one of three groups: PHiD-CV10 at 2, 4, 6 months or PCV13 at 2,4,6 months, or an investigational group of a 4-dose combination schedule of PHiD-CV10 at 1,2, and 4 months plus PCV13 at 6 months.

PREV-IX_BOOST builds on PREV-IX_COMBO to address questions not answerable by a booster trial in the general population:

The 7 month visit is the final assessment included in the PREV-IX_COMBO trial. In October 2011 the standard PCV schedule for all Indigenous babies in the NT switched from PHiD-CV10 to PCV13 at 2, 4, 6 and 18 months of age. Thus, all babies in PREV-IX_COMBO will go on to receive PCV13 at 18 months of age as a part of standard care. An alternative and innovative option is to take this opportunity to answer these questions: should PCV13 or PHiD-CV10 vaccine be the booster vaccine for infants in the three PREV-IX_COMBO groups, and at what age should the booster be given? Secondary questions: By randomising the three different primary course groups to booster dose of either PHiD-CV10 or PCV13, a number of secondary questions can be proposed. Outputs include the comparative benefit (immune and carriage correlates) of schedules such as 3+1 PCV13, 3+1 PHiD-CV10, and mixed vaccine schedules such as single dose PCV13 or single dose PHiD-CV10 boosters following alternate vaccines in the primary course, and booster options following the early and mixed 4-dose primary course. Furthermore the design will allow for an evaluation at 18 months of age, of a 12 month boost versus no boost of specific vaccine components unique to each of these vaccines. For example, a comparison of the booster effect of HiD (in PHiD-CV10) with no HiD boost (PCV13) on antibody concentration and nasopharyngeal carriage at 18 months. By combining some of these groups it will be possible to compare more subtle differences such as differences in immunogenicity of serotypes shared by the two vaccines (1,4,5,6B,7F,9V,14,18C,19F,23F) but with different carrier proteins and thus anticipated differences in immunogenicity.

PCVs in the NT: PCV7, PHiD-CV10 (Synflorix) and PCV13 (Prevenar13):

Prevention of invasive pneumococcal disease (IPD) is the primary goal of pneumococcal conjugate vaccination in infants. Effectiveness against overall IPD has generally remained high although IPD caused by non-PCV7 types has increased in some high risk groups and regions, particularly associated with serotypes 19A, 6A, and 33F. These increases have been described as a 'replacement phenomenon'. In addition there are ongoing outbreaks of IPD due to non-PCV7 types; in the NT and WA serotypes 1 and 12F account for resurgence in IPD cases in otherwise low risk groups. Effectiveness of PCVs for all-cause pneumonia and otitis media has been greatly compromised by replacement serotypes and the broad diversity of non-pneumococcal respiratory bacterial pathogens which continue to cause high rates of disease, such as non-typeable H. influenzae (NTHi). Replacement serotypes, particularly 19A(2,3) and NTHi, are the targets of new generation vaccines. In Australia two new PCVs are licensed: 10-valent pneumococcal-Haemophilus influenzae protein-D conjugate vaccine, PHiD-CV10 (Synflorix, GSK) and 13-valent PCV, PCV13 (Prevenar13, Pfizer). The two vaccines have 10 pneumococcal serotypes in common (1,4,5,6B,7F,9V,14,18C,19F,23F), however these are conjugated to different carrier proteins and immune correlates indicate potential vaccine differences in efficacy for individual serotypes. PHiD-CV10 has protein D of NTHi as the carrier for some serotypes and PCV13 is non-toxic diphtheria protein (CRM197)-conjugated, as was its precursor PCV7, and has three additional serotypes (3, 6A and 19A) but not HiD. There have been no efficacy trials that directly compare these vaccines; licensure has been based on immune correlates of protection in comparison with PCV7. Evidence of HiD efficacy has come from a single RCT in which otitis media was a primary outcome. In that trial of the original formulation (PHiD-CV11) there was ~55% efficacy for vaccine type AOM, and 35% efficacy for NTHi AOM following a 3+1 schedule.(3) This trial also demonstrated a 43% (95% Confidence Interval (CI): -17 to 72, ns) reduction in the carriage of vaccine serotypes and a 43% (95% CI: 1-67) reduction in the carriage of H. influenzae. This finding has not been replicated in later trials, partially due to very low baseline rates of NTHi carriage (<10%) and thus low power to achieve statistical significance. The PREV-IX_COMBO trial will therefore be very important in providing data on immunological correlates and carriage for different PHiD-CV10 schedules. However, an extended follow-up and comparison of booster dose (this PREV-IX_BOOST proposal) will provide further evidence for or against inclusion of PHiD-CV10 as a booster (compared to the NT standard PCV13 at 18 months).

In the NT, booster pneumococcal vaccines are recommended at 18 months of age. This is largely due to the previous schedule which included 23-valent pneumococcal polysaccharide vaccine (23PPV) as a booster dose at 18 months. A 3+1 PHiD-CV10 schedule replaced 3+1 PCV7-23PPV in 2009, and the booster age remained at 18 months. In Queensland (QLD) and in Western Australia (WA) the vaccination schedules allow for PCV13 boost at 12 months of age for high risk and Indigenous children.

At present there are 4 intra-muscular immunizations (IMIs) at 12 months of age for Indigenous infants in the Northern Territory childhood vaccination schedule. A combined booster dose vaccine (e.g. Menitorix) became available in Australia prior to commencement of first enrolment into the BOOST study. This reduces the number of IMIs at 12 months of age and provides a 'space' for PCV at 12 months. Administration of PCV booster, originally scheduled for 13 months of age, will be at 12 months of age for the trial.

Surveillance of otitis media in remote communities shows high rates of disease from weeks after birth throughout early childhood, particularly tympanic membrane perforations in the second year of life, and thus supports the need for a booster dose. Between 2008 and 2010, in PCV7-vaccinated children, mean age of tympanic membrane perforation was 18 months; for children with AOM with perforation (AOMwiP), the mean age was 13 months and for chronic suppurative OM (CSOM) 21 months. IPD cases occurring in Indigenous and non-Indigenous children less than 2 years of age for all serotypes; in 2009 there were 7 cases; in 2011 8 cases. The majority of IPD cases in children under 2 years occurred between 12 and 18 months.

In summary, the precedent of a 12 month PCV booster for Indigenous children in WA and QLD, and the high incidence of IPD and OM in the first half of the second year of life support the decision to choose a 12 month booster for this study. The mixed schedules will still allow us to compare boost versus no boost for HiD, 3,6A and 19A.

Antibody decay post-primary PCV7 to pre-booster:

Furthermore, published data(4) from the PCV7 era which show post-primary antibody levels at mean age 15 months (range 0.32 to 0.83 microg/mL for all but serotype 14) have declined almost to those detected in cord blood (range 0.3647 to 1.1797 microg/mL). The clinical implications of this decay in terms of memory response and duration of protection from mucosal infections, pneumonia and otitis media, are not known, however vaccine efficacy is lower for mucosal compared to invasive infection(5). Which vaccine for the booster dose?

Mucosal disease (OM and respiratory illness):

Culture of ear discharge from these perforations shows 60% of specimens from AOMwiP cultured NTHi and 26% cultured pneumococcus. For CSOM, these figures were 47% and 23% respectively. Serotyping identified 19A or 6A in 20% of pneumococcal isolates, which translates to 5% AOMwip and 4% CSOM specimens. NTHi is also associated with exacerbations of chronic suppurative lung disease (CSLD), or bronchiectasis, in young Indigenous children.(6) Percentage of ear discharge specimens with OM pathogens pneumococcus (Spn), 19A, NTHi, M. catarrhalis or neither Spn nor NTHi.

Evidence for efficacy of single dose PHiD-CV10 boost & inclusion in Australian PCV13 3+0 schedule:

A single dose of PHiD-CV10 might be valuable for many Australian children now receiving the 3+0 PCV13 schedule, to provide some immune protection from NTHi. Group 2 of the PREV-IX_COMBO trial receive either PCV13 at 2,4,6 months and will be randomised in this study to PCV13 (4th dose) or PHiD-CV10 (1st dose) at 12 months of age. Vesikari et al.(7) evaluated a single dose of PHiD-CV as catch-up (not booster) in 2 to 5 year old children. Following 1 dose in the 2 to 5 years group ELISA pneumococcal responses were lower than the reference group (reference group: 3 primary doses with booster at 12 to 15 months) for several serotypes. Responses following 1 dose in children 2 to 5 years of age suggested that 2 doses may be preferable. Unfortunately, HiD Geometric Mean Concentrations (GMCs) were not reported. A trial underway in Queensland will evaluate a double dose of PHiD-CV10 in preventing exacerbations of CSLD in older children. The BOOST trial in non-CSLD children will complement those data.

Invasive disease due to PCV13 serotypes 3, 6A and 19A:

In 2009, there were 89 cases of IPD in the NT population, 59 in 2010 and 114 in 2011; 25 (10%) of these 262 cases were the unique PCV13 serotypes (3, 6A and 19A) and 17(7%) of these were Indigenous, four (1.5%) were Aboriginal children < 2 years of age - about one per year (unpublished, Centre for Disease Control, NT Health).

Episodes of AOM and respiratory illness to 3 years of age:

A very high rate of clinic presentations occurs for babies and young children in remote communities. Our antibiotic trial for prevention of OM randomised infants at mean age 5 months(9,10) and recorded episodes of illness in placebo and active groups during approximately 6 months (unpublished). Around 9 episodes of primary respiratory illness or AOM (8.2 + 0.8) were recorded in notes per child year in the second 6 months of life. There are no published data for illness in the second and third years of life for this population. Whilst the BOOST study is unlikely to be sufficiently powered to detect group differences in rates of illness, these will be measured and reported.

ELIGIBILITY:
Inclusion Criteria:

* Australian Indigenous infant who was a participant in PREV-IX_COMBO trial of primary course pneumococcal conjugate vaccines, age at least 2 months post final dose of primary course. Signed informed consent.

Exclusion Criteria:

* adverse reaction to Prevenar13 or Synflorix

Ages: 9 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 261 (Actual)
Dates: Start 2013-03-12 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Immune response | At 18 months of age
  The primary outcome will be the proportion of subjects with serotype-specific antibody above the level required for protection from IPD in each study group at 18 months of age, 6 months after the booster dose. This will be determined in ELISA assays.

SECONDARY OUTCOMES:
Nasopharyngeal carriage | At 12, 18 and 36 months of age
  At baseline (12 mo), 18 and 36 months of age, the proportion of children with a any carriage of serotype 3, 6A and 19A pneumococci b any carriage of any NTHi
Otitis media | At 12, 18 and 36 months of age
  At baseline (12 mo), 18 and 36 months of age, the proportion of children with c any otitis media. d any tympanic membrane perforation

OTHER OUTCOMES:
Episodes of respiratory illness and acute otitis media | Between baseline (12 mo) and 36 months of age
  Between baseline (12 mo) and 36 months of age Episodes of respiratory illness and acute otitis media

CONTACTS AND LOCATIONS:
Overall Officials: Amanda J Leach, PhD, Principal Investigator — Menzies School of Health Research
Locations (1):
- Menzies School of Health Research, Darwin, Northern Territory, Australia

REFERENCES:
- [Background] Williams SR, Mernagh PJ, Lee MH, Tan JT. Changing epidemiology of invasive pneumococcal disease in Australian children after introduction of a 7-valent pneumococcal conjugate vaccine. Med J Aust. 2011 Feb 7;194(3):116-20. doi: 10.5694/j.1326-5377.2011.tb04192.x. PMID 21299484
- [Background] Miller E, Andrews NJ, Waight PA, Slack MP, George RC. Effectiveness of the new serotypes in the 13-valent pneumococcal conjugate vaccine. Vaccine. 2011 Nov 15;29(49):9127-31. doi: 10.1016/j.vaccine.2011.09.112. Epub 2011 Oct 5. PMID 21983361
- [Background] Weinberger DM, Malley R, Lipsitch M. Serotype replacement in disease after pneumococcal vaccination. Lancet. 2011 Dec 3;378(9807):1962-73. doi: 10.1016/S0140-6736(10)62225-8. Epub 2011 Apr 12. PMID 21492929
- [Background] Leach AJ, Morris PS, Mackenzie G, McDonnell J, Balloch A, Carapetis J, Tang M. Immunogenicity for 16 serotypes of a unique schedule of pneumococcal vaccines in a high-risk population. Vaccine. 2008 Jul 23;26(31):3885-91. doi: 10.1016/j.vaccine.2008.05.012. Epub 2008 May 27. PMID 18562052
- [Background] Black S, Shinefield H, Fireman B, Lewis E, Ray P, Hansen JR, Elvin L, Ensor KM, Hackell J, Siber G, Malinoski F, Madore D, Chang I, Kohberger R, Watson W, Austrian R, Edwards K. Efficacy, safety and immunogenicity of heptavalent pneumococcal conjugate vaccine in children. Northern California Kaiser Permanente Vaccine Study Center Group. Pediatr Infect Dis J. 2000 Mar;19(3):187-95. doi: 10.1097/00006454-200003000-00003. PMID 10749457
- [Background] Hare KM, Grimwood K, Leach AJ, Smith-Vaughan H, Torzillo PJ, Morris PS, Chang AB. Respiratory bacterial pathogens in the nasopharynx and lower airways of Australian indigenous children with bronchiectasis. J Pediatr. 2010 Dec;157(6):1001-5. doi: 10.1016/j.jpeds.2010.06.002. Epub 2010 Jul 24. PMID 20656297
- [Background] Vesikari T, Karvonen A, Korhonen T, Karppa T, Sadeharju K, Fanic A, Dieussaert I, Schuerman L. Immunogenicity of 10-valent pneumococcal nontypeable Haemophilus Influenzae Protein D Conjugate Vaccine when administered as catch-up vaccination to children 7 months to 5 years of age. Pediatr Infect Dis J. 2011 Aug;30(8):e130-41. doi: 10.1097/INF.0b013e31821d1790. PMID 21540760
- [Background] Clucas DB, Carville KS, Connors C, Currie BJ, Carapetis JR, Andrews RM. Disease burden and health-care clinic attendances for young children in remote aboriginal communities of northern Australia. Bull World Health Organ. 2008 Apr;86(4):275-81. doi: 10.2471/blt.07.043034. PMID 18438516
- [Background] Leach AJ, Morris PS, Mathews JD; Chronic Otitis Media Intervention Trial - One (COMIT1) group. Compared to placebo, long-term antibiotics resolve otitis media with effusion (OME) and prevent acute otitis media with perforation (AOMwiP) in a high-risk population: a randomized controlled trial. BMC Pediatr. 2008 Jun 2;8:23. doi: 10.1186/1471-2431-8-23. PMID 18513453
- [Background] Simell B, Nurkka A, Lahdenkari M, Givon-Lavi N, Kayhty H, Dagan R, Jokinen J. Association of serotype-specific antibody concentrations and functional antibody titers with subsequent pneumococcal carriage in toddlers immunized with a 9-valent pneumococcal conjugate vaccine. Clin Vaccine Immunol. 2012 Jan;19(1):96-9. doi: 10.1128/CVI.05369-11. Epub 2011 Nov 9. PMID 22072724
- [Background] Leach AJ, Morris PS, McCallum GB, Wilson CA, Stubbs L, Beissbarth J, Jacups S, Hare K, Smith-Vaughan HC. Emerging pneumococcal carriage serotypes in a high-risk population receiving universal 7-valent pneumococcal conjugate vaccine and 23-valent polysaccharide vaccine since 2001. BMC Infect Dis. 2009 Aug 4;9:121. doi: 10.1186/1471-2334-9-121. PMID 19650933
- [Background] Prymula R, Kriz P, Kaliskova E, Pascal T, Poolman J, Schuerman L. Effect of vaccination with pneumococcal capsular polysaccharides conjugated to Haemophilus influenzae-derived protein D on nasopharyngeal carriage of Streptococcus pneumoniae and H. influenzae in children under 2 years of age. Vaccine. 2009 Dec 10;28(1):71-8. doi: 10.1016/j.vaccine.2009.09.113. Epub 2009 Oct 8. PMID 19818722
- [Background] Prymula R, Peeters P, Chrobok V, Kriz P, Novakova E, Kaliskova E, Kohl I, Lommel P, Poolman J, Prieels JP, Schuerman L. Pneumococcal capsular polysaccharides conjugated to protein D for prevention of acute otitis media caused by both Streptococcus pneumoniae and non-typable Haemophilus influenzae: a randomised double-blind efficacy study. Lancet. 2006 Mar 4;367(9512):740-8. doi: 10.1016/S0140-6736(06)68304-9. PMID 16517274
- [Derived] Leach AJ, Wilson N, Arrowsmith B, Beissbarth J, Mulholland K, Santosham M, Torzillo PJ, McIntyre P, Smith-Vaughan H, Skull SA, Oguoma VM, Chatfield MD, Lehmann D, Brennan-Jones CG, Binks MJ, Licciardi PV, Andrews RM, Snelling T, Krause V, Carapetis J, Chang AB, Morris PS. Hearing loss in Australian First Nations children at 6-monthly assessments from age 12 to 36 months: Secondary outcomes from randomised controlled trials of novel pneumococcal conjugate vaccine schedules. PLoS Med. 2024 Jun 3;21(6):e1004375. doi: 10.1371/journal.pmed.1004375. eCollection 2024 Jun. PMID 38829821
- [Derived] Leach AJ, Wilson N, Arrowsmith B, Beissbarth J, Mulholland EK, Santosham M, Torzillo PJ, McIntyre P, Smith-Vaughan H, Chatfield MD, Lehmann D, Binks M, Chang AB, Carapetis J, Krause V, Andrews R, Snelling T, Skull SA, Licciardi PV, Oguoma VM, Morris PS. Immunogenicity, otitis media, hearing impairment, and nasopharyngeal carriage 6-months after 13-valent or ten-valent booster pneumococcal conjugate vaccines, stratified by mixed priming schedules: PREVIX_COMBO and PREVIX_BOOST randomised controlled trials. Lancet Infect Dis. 2022 Sep;22(9):1374-1387. doi: 10.1016/S1473-3099(22)00272-9. Epub 2022 Jun 27. PMID 35772449
- [Derived] Oguoma VM, Wilson N, Mulholland K, Santosham M, Torzillo P, McIntyre P, Smith-Vaughan H, Balloch A, Chatfield M, Lehmann D, Binks MJ, Chang A, Carapetis J, Krause V, Andrews R, Snelling T, Licciardi P, Morris P, Leach AJ. 10-Valent pneumococcal non-typeable H. influenzae protein D conjugate vaccine (PHiD-CV10) versus 13-valent pneumococcal conjugate vaccine (PCV13) as a booster dose to broaden and strengthen protection from otitis media (PREVIX_BOOST) in Australian Aboriginal children: study protocol for a randomised controlled trial. BMJ Open. 2020 May 24;10(5):e033511. doi: 10.1136/bmjopen-2019-033511. PMID 32448790